CLINICAL TRIAL: NCT00795977
Title: Phase I/II Study on Intratumor Dendritic Cell Injection Immunotherapy Using Immature Dendritic Cells With S Pyogenes Preparation (OK-432) for Patients With Resectable Pancreatic Cancer
Brief Title: Preoperative Intratumor Dendritic Cells Injection Immunotherapy for Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fukushima Medical University (Other)
Responsible Party: Principal Investigator, Akira Kenjo, Department of Surgery I, Fukushima Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 198
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Pancreatic Cancer
Keywords: preoperative; intratumor; dendritic cells; pancreatic cancer; OK-432
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Picibanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dendritic cells (Experimental)
  Interventions: Biological: dendritic cells, OK-432

INTERVENTIONS:
Biological: dendritic cells, OK-432 — Single Group Assignment

SUMMARY:
The purpose of this study is to confirm safety and immunological responses of Preoperative intratumor dendritic cells injection immunotherapy using immature dendritic cells with S pyogenes Preparation (OK-432) for patients with resectable pancreatic cancer for pancreatic cancer patients.

DETAILED DESCRIPTION:
The prognosis of pancreatic cancer is extremely poor even with extensive surgery, and development of new treatment modalities is much-expected for cure of this disease. Dendritic cells (DCs) immunotherapy is expected favorable outcome when it is approached directly to the cancer tissue. To evaluate safety and immunological responses, we conducted a phase I/II study of intra-tumor DCs immunotherapy for pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Resectable pancreatic cancer without distant metastasis:

1. ECOG performance status 0-2
2. Laboratory values as follows 3,500/mm3 <WBC<12000/mm3 Platelet count>100,000/mm3 T-Bil<2.0mg/dl BUN<25mg/dl, Creatinin<1.5mg/dl, 24h Ccr>50ml/min Normal ECG
3. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breast-feeder
3. Active or uncontrolled infection
4. Active or uncontrolled other malignancy
5. Steroids or immunosuppressing agent dependant status
6. Interstitial pneumonia
7. Decision of unsuitableness by principal investigator or physician-in-charge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
To establish the maximally tolerated dose (MTD) and dose limiting toxicities (DLT) of intratumoral autologous dendritic cell vaccination in combination with OK-432 | 2 years

SECONDARY OUTCOMES:
To determine the overall response rate for this regimen as determined by overall and disease-free survival. | 2 years
To evaluate the immune response of patients treated with this regimen based on the presence and characterization of tumor-infiltrating white blood cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitsukazu Gotoh, MD & PhD, Study Chair — Fukushima Medical University, Department of Surgery 1
Locations (1):
- Fukushima Medical University Hospital, Fukushima, Japan

REFERENCES:
- [Background] Kanzaki N, Terashima M, Kashimura S, Hoshino M, Ohtani S, Matsuyama S, Hoshino Y, Kogure M, Oshibe I, Endo H, Saito T, Yaginuma H, Gotoh M, Ohto H. Understanding the response of dendritic cells to activation by streptococcal preparation OK-432. Anticancer Res. 2005 Nov-Dec;25(6B):4231-8. PMID 16309221
- [Background] Takekuni K, Sakon M, Kishimoto S, Amano M, Sekimoto M, Aoki T, Oosato H, Dohno K, Umeshita K, Gotoh M, Monden T, Monden M. [A patient with unresectable cancer of pancreas head, effectively treated by a local injection of the mixture of OK-432, fibrinogen and thrombin]. Gan To Kagaku Ryoho. 1996 Sep;23(11):1621-3. Japanese. PMID 8854822
- [Background] Okamoto M, Furuichi S, Nishioka Y, Oshikawa T, Tano T, Ahmed SU, Takeda K, Akira S, Ryoma Y, Moriya Y, Saito M, Sone S, Sato M. Expression of toll-like receptor 4 on dendritic cells is significant for anticancer effect of dendritic cell-based immunotherapy in combination with an active component of OK-432, a streptococcal preparation. Cancer Res. 2004 Aug 1;64(15):5461-70. doi: 10.1158/0008-5472.CAN-03-4005. PMID 15289356
- [Background] Oshikawa T, Okamoto M, Ahmed SU, Tano T, Yoshida H, Sato M. [Anti-cancer effect of an intratumoral injection of dendritic cells expressing TLR4 in combination with an active component of OK-432 in TLR4-deficient mice]. Gan To Kagaku Ryoho. 2004 Oct;31(11):1770-2. Japanese. PMID 15553710